CLINICAL TRIAL: NCT01974687
Title: A Phase I/IIa Study Assessing Single and Multiple Doses of IDX21437 in Healthy and HCV-Infected Subjects
Brief Title: Single and Multiple Dose Study of Uprifosbuvir (MK-3682/IDX21437) in Healthy and Hepatitis C Virus (HCV)-Infected Participants (MK-3682-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3682-001; U1111-1149-5611 (Other: Universal Trial Number (UTN)); IDX-04B-001 (Other: Idenix Protocol Number); 2013-004043-23 (EudraCT Number); MK-3682-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C virus; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — uprifosbuvir; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A: Healthy (Experimental): Healthy participants will receive sequentially higher doses of uprifosbuvir (10 mg - 300 mg) capsules or matching placebo capsules once daily (QD) on Day 1 (Cohorts 1a-3a, 5a), Days 1 and 7 (Cohort 4a), or Day 1 - Day 7 (Cohort 6a). Dosing of next cohort will be based on review of available safety and PK data. Dosing will occur under fasted conditions with the exception of Cohort 4a, in which drug administration will occur under both fasted and fed conditions.
  Interventions: Drug: Uprifosbuvir; Drug: Placebo
- Group B: GT1 HCV-infected, treatment naive on Day 1 (Experimental): HCV GT1 participants with no prior direct-acting antiviral (DAA) exposure will receive a single dose of uprifosbuvir (10 mg - 300 mg) for 1 day across sequential dose cohorts. Dosing will commence following review of available safety and PK data from respective dose cohorts in Group A. All dosing will occur under fasted conditions.
  Interventions: Drug: Uprifosbuvir
- Group C: GT1 HCV-infected on Days 1-7 (Experimental): HCV GT1 participants will receive uprifosbuvir (50 mg - 400 mg in capsules or 300 mg or 450 mg in tablets) or matching placebo capsules QD for 7 days. Dosing will commence following review of available safety and PK data of Group A. Fed vs. fasted dosing will be dependent on food effect results from Group A.
  Interventions: Drug: Uprifosbuvir; Drug: Placebo
- Group D: GT2 through GT6 HCV-infected on Days 1-7 (Experimental): HCV GT2 - GT6 participants will receive uprifosbuvir (50 mg - 300 mg) capsules QD for 7 days. Dosing will commence following review of available safety and PK data from Group A. Fed vs. fasted dosing will be dependent on food effect results from Group A.
  Interventions: Drug: Uprifosbuvir
- Group E: GT1 HCV-infected on Days 1-7, mild hepatic impairment (Experimental): HCV GT1 participants with mildly impaired hepatic function will receive uprifosbuvir (150 mg - 450 mg) capsules QD for 1 or 7 days. Dosing of subsequent cohorts will be based on review of available safety and PK data. Fed vs. fasted dosing will be dependent on food effect results from Group A.
  Interventions: Drug: Uprifosbuvir
- Group F: GT1 HCV-infected on Days 1-7, + Itraconazole (Experimental): HCV GT1 participants will receive itraconazole 200 mg twice daily (BID) on Day -5 and itraconazole 200 mg QD from Day -4 to Day 11. Participants will also be co-administered uprifosbuvir 300 mg from Day 1 to Day 7.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Uprifosbuvir — Uprifosbuvir 5 mg, 25 mg, or 50 mg capsule, or 150 mg tablet, administered by mouth.
  Other Names: MK-3682/IDX21437
  Arms: Group A: Healthy; Group B: GT1 HCV-infected, treatment naive on Day 1; Group C: GT1 HCV-infected on Days 1-7; Group D: GT2 through GT6 HCV-infected on Days 1-7; Group E: GT1 HCV-infected on Days 1-7, mild hepatic impairment
Drug: Placebo — Matching placebo to uprifosbuvir capsule administered by mouth.
  Arms: Group A: Healthy; Group C: GT1 HCV-infected on Days 1-7
Drug: Itraconazole — Itraconazole is supplied as 10 mg/mL oral solution or 100 mg capsules administered by mouth.
  Other Names: Sporanox®
  Arms: Group F: GT1 HCV-infected on Days 1-7, + Itraconazole

SUMMARY:
This is a multi-part study to evaluate the safety, tolerability, and pharmacokinetics (PK) of uprifosbuvir (MK-3682/IDX21437) in healthy participants and in participants infected with Hepatitis C virus (HCV) genotype (GT)1-GT6. The effect of food on the PK of uprifosbuvir will be evaluated. The antiviral activity of uprifosbuvir will also be assessed in HCV-infected participants.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* of childbearing potential must have agreed to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of the study drug
* must not have consumed grapefruit or grapefruit juice within 7 days of Day -1 and throughout the study

HCV Participants:

* documented clinical history compatible with chronic hepatitis C.
* have not received direct-acting antiviral treatment for hepatitis C infection
* has HCV Genotype 1, 2, 3, 4, 5 or 6

Exclusion Criteria:

All Participants:

* pregnant or breastfeeding
* co-infected with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV).
* decompensated liver disease
* other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2015-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, the Group D part of the study allowed to randomize Genotype 2, 3, 4, 5 and 6 Hepatitis C Virus (HCV)-infected participants, however, only Genotype 2 and 3 HCV-infected participants were enrolled.
Groups:
- Group A: Uprifosbuvir 10 mg (Cohort 1a): Participants were administered a single dose of uprifosbuvir (MK-3682/IDX21437) 10 mg as oral capsules under fasted conditions.
- Group A: Uprifosbuvir 25 mg (Cohort 2a); Group B: Uprifosbuvir 25 mg (Cohort 2b): Participants were administered a single dose of uprifosbuvir 25 mg as oral capsules under fasted conditions.
- Group A: Uprifosbuvir 150 mg (Cohort 4a): Participants were administered single doses of uprifosbuvir 150 mg as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods.
- Group A: Uprifosbuvir 300 mg (Cohort 5a); Group B: Uprifosbuvir 300 mg (Cohort 5b): Participants were administered a single dose of uprifosbuvir 300 mg as oral capsules under fasted conditions.
- Group A: Placebo (Cohort 6a): Participants were administered single doses of uprifosbuvir-matching placebo oral capsules once daily for 7 days under fasted conditions.
- Group A: Uprifosbuvir 300 mg (Cohort 6a); Groups C & D: Uprifosbuvir 300 mg (Capsule); Group E: Uprifosbuvir 300 mg (Cohort 2e): Participants were administered single doses of uprifosbuvir 300 mg as oral capsules once daily for 7 days under fasted conditions.
- Group B: Uprifosbuvir 10 mg (Cohort 1b): Participants were administered a single dose of uprifosbuvir 10 mg as oral capsules under fasted conditions.
- Group B: Uprifosbuvir 50 mg (Cohort 3b); Group A: Uprifosbuvir 50 mg (Cohort 3a): Participants were administered a single dose of uprifosbuvir 50 mg as oral capsules under fasted conditions.
- Group B: Uprifosbuvir 150 mg (Cohort 4b); Group E: Uprifosbuvir 150 mg (Cohort 1e): Participants were administered a single dose of uprifosbuvir 150 mg as oral capsules under fasted conditions.
- Groups C & D: Uprifosbuvir 50 mg (Capsule): Participants were administered single doses of uprifosbuvir 50 mg as oral capsules once daily for 7 days under fasted conditions.
- Groups C & D: Uprifosbuvir 150 mg (Capsule): Participants were administered single doses of uprifosbuvir 150 mg as oral capsules once daily for 7 days under fasted conditions.
- Groups C & D: Uprifosbuvir 250 mg (Capsule): Participants were administered single doses of uprifosbuvir 250 mg as oral capsules once daily for 7 days under fasted conditions.
- Groups C & D: Uprifosbuvir 400 mg (Capsule): Participants were administered single doses of uprifosbuvir 400 mg as oral capsules once daily for 7 days under fasted conditions.
- Groups C & D: Uprifosbuvir 300 mg (Tablet): Participants were administered single doses of uprifosbuvir 300 mg as oral tablets once daily for 7 days under fasted conditions.
- Groups C & D: Uprifosbuvir 450 mg (Tablet); Group E: Uprifosbuvir 450 mg (Cohort 3e): Participants were administered single doses of uprifosbuvir 450 mg as oral tablets once daily for 7 days under fasted conditions.
- Groups C & D: Placebo (Pooled): Participants were administered single doses of uprifosbuvir-matching placebo as oral capsules once daily for 7 days under fasted conditions.
- Group F: Uprifosbuvir 300 mg (Tablet): Participants were administered single doses of uprifosbuvir 300 mg as oral tablets once daily for 7 days under fasted conditions. Participants were also administered itraconazole 200 mg twice daily as oral solution on Day -5 and 200 mg once daily from Day -4 to Day 11.
- Group A: Placebo (Cohorts 1a-5a - Pooled): Participants were administered a single dose of uprifosbuvir-matching placebo as oral capsules under fasted conditions (Cohorts 1a, 2a, 3a, 5a); Participants were administered single doses of uprifosbuvir-matching placebo as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods (Cohort 4a).
Period: Overall Study
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Placebo (Cohort 6a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Placebo (Cohorts 1a-5a - Pooled)
Started | 6 | 6 | 6 | 6 | 2 | 6 | 3 | 3 | 3 | 3 | 3 | 13 | 13 | 10 | 19 | 9 | 9 | 11 | 9 | 3 | 3 | 8 | 8 | 6 | 10
Treated | 6 | 6 | 6 | 6 | 2 | 6 | 3 | 3 | 3 | 3 | 3 | 11 (2 participants discontinued prior to receiving study drug) | 10 (3 participants discontinued prior to receiving study drug) | 8 (2 participants discontinued prior to receiving study drug) | 18 (1 participant discontinued prior to receiving study drug) | 8 (1 participant discontinued prior to receiving study drug) | 8 (1 participant discontinued prior to receiving study drug) | 8 (3 participants discontinued prior to receiving study drug) | 9 | 3 | 3 | 8 | 8 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 2 | 6 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all participants who received at least one dose of study drug.
Groups:
- Group A: Placebo (Cohort 1a-Cohort 5a - Pooled): Participants were administered a single dose of uprifosbuvir-matching placebo as oral capsules under fasted conditions (Cohorts 1a, 2a, 3a, 5a); Participants were administered single doses of uprifosbuvir-matching placebo as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods (Cohort 4a).
- Group A: Uprifosbuvir 10 mg (Cohort 1a); Group B: Uprifosbuvir 10 mg (Cohort 1b): Participants were administered a single dose of uprifosbuvir 10 mg as oral capsules under fasted conditions.
- Total: Total of all reporting groups
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Placebo (Cohort 6a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 2 | 6 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8 | 6 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 6 | 6 | 6 | 2 | 6 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8 | 6 | 165
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (7.72) | 29.2 (7.36) | 33.3 (15.06) | 35.5 (11.76) | 35.2 (9.87) | 36.0 (2.83) | 35.3 (12.69) | 37.0 (9.54) | 42.3 (7.23) | 46.7 (4.16) | 43.3 (5.69) | 41.3 (8.96) | 41.2 (10.68) | 42.7 (10.37) | 44.3 (8.63) | 40.1 (11.69) | 43.3 (8.45) | 40.5 (11.70) | 40.5 (8.94) | 43.7 (7.68) | 57.0 (4.36) | 56.3 (3.06) | 49.1 (8.04) | 43.1 (12.54) | 31.3 (11.60) | 40.47 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 5 | 4 | 0 | 4 | 0 | 0 | 1 | 2 | 1 | 5 | 0 | 5 | 5 | 3 | 5 | 4 | 3 | 0 | 0 | 1 | 6 | 3 | 67
  Male | 6 | 2 | 4 | 1 | 2 | 2 | 2 | 3 | 3 | 2 | 1 | 2 | 6 | 10 | 3 | 13 | 5 | 3 | 4 | 6 | 3 | 3 | 7 | 2 | 3 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug, and that does not necessarily have a causal relationship with the study drug(s). An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug(s), whether or not related to study drug(s). The percentage of participants who experienced at least one AE is presented.
Time Frame: Up to 42 days
Population: Safety Population: all participants who received at least one dose of the study drug
Measure: Number; unit: Percentage of Participants
Groups:
- Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed): Participants were administered single doses of uprifosbuvir 150 mg as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods.
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group A: Placebo (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8
Percentage of Participants | 50.0 | 0.0 | 33.3 | 33.3 | 66.7 | 50.0 | 33.3 | 50.0 | 33.3 | 66.7 | 33.3 | 66.7 | 66.7 | 72.7 | 70.0 | 87.5 | 44.4 | 62.5 | 75.0 | 62.5 | 66.7 | 0.0 | 100.0 | 62.5 | 37.5

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Serious AE (SAE)
Description: An SAE was defined as any untoward medical occurrence that at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. The percentage of participants who experienced at least one SAE is presented.
Time Frame: Up to 42 days
Population: Safety Population: all participants who received at least one dose of the study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group A: Placebo (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants Who Experienced a Treatment-emergent Dose-limiting Toxicity (DLT)
Description: A DLT was defined as any of the following events: Any SAE considered by the investigator to be at least reasonably or possibly related to study drug; Any Grade 3 clinical AE considered by the investigator to be at least reasonably or possibly related to study drug; Any Grade 3 confirmed laboratory abnormalities considered by the investigator to be at least reasonably or possibly related to study drug, except for asymptomatic Grade ¾ cholesterol and triglyceride; Any clinical or laboratory AE of any intensity that is considered by the investigator to be at least reasonably or possibly related to study drug that necessitates permanent discontinuation of study drug; Confirmed increase in QT interval corrected for heart rate using Fridericia's (QTcF) formula ≥60 msec over Baseline or an absolute QTcF ≥500 msec.
Time Frame: Up to 13 days
Population: Safety Population: all participants who received at least one dose of the study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group A: Placebo (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Grade 1, 2, 3, 4 or 5 Laboratory Abnormality
Description: Laboratory abnormalities were graded using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Treatment-emergent AEs (TEAEs)were graded as: Grade 1: Mild TEAE as Worst Severity; Grade 2: Moderate TEAE as Worst Severity; Grade 3: Severe TEAE as Worst Severity; Grade 4: Potentially Life-Threatening TEAE as Worst Severity; Grade 5: TEAE Leading to Death. The percentage of participants who experienced at least one Grade 1, 2, 3, 4 or 5 laboratory abnormality is presented.
Time Frame: Up to 42 days
Population: Safety Population: all participants who received at least one dose of the study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group A: Placebo (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8
Percentage of Participants
  Grade 1 | 50.00 | 0.0 | 16.7 | 16.7 | 50.0 | 33.3 | 33.3 | 50.0 | 0.0 | 66.7 | 33.3 | 66.7 | 66.7 | 45.5 | 60.0 | 37.5 | 33.3 | 0.0 | 37.5 | 25.0 | 33.3 | 0.0 | 100.0 | 12.5 | 0.0
  Grade 2 | 0.0 | 0.0 | 16.7 | 16.7 | 16.7 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 18.2 | 0.0 | 50.0 | 5.6 | 62.5 | 37.5 | 25.0 | 33.3 | 0.0 | 0.0 | 37.5 | 37.5
  Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 10.0 | 0.0 | 5.6 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Grade 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to a Treatment-emergent AE
Description: The percentage of participants who discontinued study drug due to an AE is presented.
Time Frame: Up to 14 days
Population: Safety Population: all participants who received at least one dose of the study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo (Cohort 1a-Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (Fasted and Fed) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group A: Placebo (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 8 | 18 | 8 | 8 | 8 | 9 | 3 | 3 | 8 | 8
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Area Under the Plasma Drug Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: Pharmacokinetics (PK) Population: a subpopulation of the per-protocol population, selecting all participants exposed to uprifosbuvir who had available and evaluable data (e.g., excluding deviations and/or other events that could have an impact on the PK analysis).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Groups:
- Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted): Participants were administered single doses of uprifosbuvir 150 mg as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods.
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*umol/L | 0.0410 (32.7) | 0.0837 (27.9) | 1.67 (62.7) | 2.78 (37.7) | 0.246 (63.2)

7. Primary Outcome: AUC0-t of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: PK Population: a subpopulation of the per-protocol population, selecting all participants exposed to uprifosbuvir who had available and evaluable data (e.g., excluding deviations and/or other events that could have an impact on the PK analysis).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Groups:
- Group A: Uprifosbuvir 150 mg (Cohort 4a Fed): Participants were administered single doses of uprifosbuvir 150 mg as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods.
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
h*umol/L | 1.05 (48.5)

8. Primary Outcome: AUC0-t of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
h*umol/L
  Day 1 | 3.62 (34.0)
  Day 7 | 3.77 (21.7)

9. Primary Outcome: AUC0-t of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
h*umol/L | 0.0640 (39.8) | 0.228 (49.1) | 0.341 (20.4) | 1.17 (NA) — Not calculated | 1.39 (35.4)

10. Primary Outcome: AUC0-t of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
h*umol/L
  Day 1 | 0.394 (51.4) | 1.01 (52.9) | 2.80 (45.4) | 5.54 (40.1)
  Day 7 | 0.347 (36.2) | 0.935 (36.7) | 2.42 (46.8) | 4.59 (22.1)

11. Primary Outcome: AUC0-t of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Groups:
- Group C: Uprifosbuvir 300 mg (Tablet): Participants were administered single doses of uprifosbuvir 300 mg as oral tablets once daily for 7 days under fasted conditions.
- Group C: Uprifosbuvir 450 mg (Tablet): Participants were administered single doses of uprifosbuvir 450 mg as oral tablets once daily for 7 days under fasted conditions.
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
h*umol/L
  Day 1 | 2.00 (51.7) | 3.11 (45.0)
  Day 7 | 1.82 (43.9) | 2.88 (30.4)

12. Primary Outcome: AUC0-t of Uprifosbuvir After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
h*umol/L | 1.05 (NA) — Not calculated

13. Primary Outcome: AUC0-t of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
h*umol/L
  Day 1 | 3.19 (32.8) | 4.21 (35.2)
  Day 7 | 2.31 (31.8) | 3.51 (23.2)

14. Primary Outcome: AUC0-t of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
h*umol/L
  Day 1 | 10.6 (44.0)
  Day 7 | 9.39 (46.1)

15. Primary Outcome: Maximum (Peak) Observed Plasma Drug Concentration (Cmax) of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: Maximum observed plasma drug concentration was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nmol/L | 29.6 (45.3) | 47.7 (54.4) | 1120 (47.8) | 1530 (53.6) | 119 (89.2)

16. Primary Outcome: Cmax of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
nmol/L | 293 (63.0)

17. Primary Outcome: Cmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
nmol/L
  Day 1 | 2300 (26.6)
  Day 7 | 2320 (19.9)

18. Primary Outcome: Cmax of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
nmol/L | 43.6 (60.7) | 122 (26.4) | 168 (11.4) | 510 (NA) — Not calculated | 667 (15.3)

19. Primary Outcome: Cmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: Maximum observed plasma drug concentration was obtained. All participants were fasted.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
nmol/L
  Day 1 | 286 (77.1) | 524 (80.1) | 1360 (55.5) | 2320 (50.2)
  Day 7 | 199 (45.6) | 587 (34.9) | 1200 (59.4) | 2490 (25.7)

20. Primary Outcome: Cmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
nmol/L
  Day 1 | 618 (45.2) | 778 (29.7)
  Day 7 | 537 (56.4) | 717 (47.2)

21. Primary Outcome: Cmax of Uprifosbuvir After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
nmol/L | 613 (NA) — Not calculated

22. Primary Outcome: Cmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
nmol/L
  Day 1 | 1440 (35.9) | 1090 (34.4)
  Day 7 | 1550 (47.5) | 929 (26.6)

23. Primary Outcome: Cmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
nmol/L
  Day 1 | 2140 (39.4)
  Day 7 | 1910 (42.6)

24. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: Time to maximum plasma concentration was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 0.80 (32.7) [0.50 to 1.05] | 1.00 (27.9) [0.50 to 3.00] | 0.76 (62.7) [0.50 to 2.00] | 0.50 (37.7) [0.50 to 2.00] | 1.00 (63.2) [0.50 to 1.00]

25. Primary Outcome: Tmax of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
hours | 3.04 (47.8) [3.00 to 4.05]

26. Primary Outcome: Tmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
hours
  Day 1 | 0.75 (26.6) [0.50 to 1.00]
  Day 7 | 0.50 (19.9) [0.50 to 2.03]

27. Primary Outcome: Tmax of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-infected Participants (Group B)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
hours | 0.50 (39.8) [0.50 to 1.00] | 1.00 (49.1) [0.53 to 1.00] | 1.00 (20.4) [0.68 to 1.00] | 0.76 (NA) [0.52 to 1.00] | 1.00 (35.4) [0.50 to 1.08]

28. Primary Outcome: Tmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-infected Participants (Groups C and D)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
hours
  Day 1 | 0.85 (51.4) [0.50 to 2.03] | 0.50 (52.9) [0.50 to 2.00] | 1.00 (45.4) [0.50 to 4.00] | 0.50 (40.1) [0.50 to 2.00]
  Day 7 | 0.97 (36.2) [0.50 to 1.00] | 0.50 (36.7) [0.50 to 1.00] | 0.50 (46.8) [0.48 to 3.00] | 0.50 (22.1) [0.50 to 3.00]

29. Primary Outcome: Tmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-infected Participants (Group C)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
hours
  Day 1 | 1.00 (51.7) [0.50 to 4.00] | 2.00 (45.0) [0.50 to 3.00]
  Day 7 | 0.50 (43.9) [0.50 to 3.00] | 0.50 (30.4) [0.50 to 3.00]

30. Primary Outcome: Tmax of Uprifosbuvir After Singe Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
hours | 0.75 (NA) [0.50 to 1.00]

31. Primary Outcome: Tmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: AUC0-t was calculated using linear log trapezoidal summation from time zero to last measurable concentration.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
hours
  Day 1 | 1.00 (32.8) [0.50 to 3.00] | 1.00 (35.2) [0.50 to 2.00]
  Day 7 | 1.00 (31.8) [0.50 to 1.00] | 1.00 (23.2) [0.50 to 2.00]

32. Primary Outcome: Tmax of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-infected Participants, With Itraconazole (Group F)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
hours
  Day 1 | 2.00 (44.0) [1.00 to 3.00]
  Day 7 | 1.00 (46.1) [1.00 to 3.00]

33. Primary Outcome: Observed Terminal Half-Life (t1/2) of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 0.839 (27.3) | 0.872 (33.7) | 1.05 (25.0) | 1.13 (31.6) | 0.979 (36.6)

34. Primary Outcome: t1/2 of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
hours | 1.63 (31.9)

35. Primary Outcome: t1/2 of Uprifosbuvir After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-infected Participants (Group B)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
hours | 1.36 (52.7) | 0.926 (34.5) | 1.09 (32.5) | 1.11 (NA) — Not calculated | 1.59 (1.7)

36. Primary Outcome: t1/2 of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-infected Participants (Groups C and D)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
hours | 1.04 (25.1) | 1.11 (22.5) | 154. (34.0) | 2.58 (40.3)

37. Primary Outcome: t1/2 of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-infected Participants (Group C)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
hours | 2.50 (55.9) | 3.64 (54.8)

38. Primary Outcome: t1/2 of Uprifosbuvir After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
hours | 1.16 (NA) — Not calculated

39. Primary Outcome: t1/2 of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
hours | 1.18 (27.2) | 2.38 (34.3)

40. Primary Outcome: t1/2 of Uprifosbuvir After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-infected Participants, With Itraconazole (Group F)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
hours | 4.30 (52.8)

41. Primary Outcome: AUC0-inf of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: Area under the drug concentration-time curve from time zero to infinity for M6, a metabolite of uprifosbuvir, estimated as AUC0-t + Cest/λz, where λz is the terminal elimination rate constant, calculated for the first dose only. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*umol/L | 1.68 (47.4) | 5.01 (27.2) | 19.8 (12.7) | 29.7 (32.1) | 8.77 (8.4)

42. Primary Outcome: AUC0-inf of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: Area under the drug concentration-time curve from time zero to infinity estimated as AUC0-t + Cest/λz, where λz is the terminal elimination rate constant, calculated for the first dose only.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
h*umol/L | 17.9 (13.4)

43. Primary Outcome: AUC0-inf of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: as for outcome 42
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
h*umol/L
  Day 1 | 15.1 (16.5)
  Day 7 | 20.6 (17.9)

44. Primary Outcome: AUC0-inf of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: as for outcome 42
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
h*umol/L | 2.26 (22.3) | 5.78 (4.7) | 7.31 (11.1) | 17.5 (NA) — Not calculated | 33.4 (37.0)

45. Primary Outcome: AUC0-inf of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: as for outcome 42
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
h*umol/L
  Day 1 | 4.74 (37.6) | 8.94 (20.2) | 14.4 (20.8) | 19.4 (11.1)
  Day 7 | 7.12 (37.6) | 12.2 (18.9) | 19.0 (16.3) | 24.4 (7.2)

46. Primary Outcome: AUC0-inf of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: as for outcome 42
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
h*umol/L
  Day 1 | 14.7 (36.6) | 16.1 (23.5)
  Day 7 | 21.4 (26.7) | 24.7 (22.5)

47. Primary Outcome: AUC0-inf of M6 After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: as for outcome 42
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
h*umol/L | 1.05 (NA) — Not calculated

48. Primary Outcome: AUC0-inf of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: as for outcome 42
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
h*umol/L
  Day 1 | 13.4 (22.3) | 18.4 (17.0)
  Day 7 | 17.5 (23.5) | 26.1 (26.5)

49. Primary Outcome: AUC0-inf of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: as for outcome 42
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*umol/L
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
h*umol/L
  Day 1 | 13.2 (32.0)
  Day 7 | 23.8 (37.0)

50. Primary Outcome: Cmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: Maximum observed plasma drug concentration was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nmol/L | 63.2 (19.8) | 146 (13.6) | 758 (28.2) | 1190 (16.6) | 283 (14.7)

51. Primary Outcome: Cmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
nmol/L | 509 (8.4)

52. Primary Outcome: Cmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
nmol/L
  Day 1 | 1310 (7.5)
  Day 7 | 1630 (14.9)

53. Primary Outcome: Cmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
nmol/L | 55.0 (15.0) | 170 (7.2) | 279 (5.2) | 710 (NA) — Not calculated | 1210 (33.8)

54. Primary Outcome: Cmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
nmol/L
  Day 1 | 298 (34.2) | 641 (7.6) | 1130 (22.7) | 1560 (18.9)
  Day 7 | 471 (33.7) | 931 (14.4) | 1420 (15.3) | 1760 (10.4)

55. Primary Outcome: Cmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
nmol/L
  Day 1 | 1010 (31.5) | 1210 (21.9)
  Day 7 | 1420 (23.2) | 1680 (21.5)

56. Primary Outcome: Cmax of M6 After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
nmol/L | 597 (NA) — Not calculated

57. Primary Outcome: Cmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
nmol/L
  Day 1 | 1100 (11.5) | 1180 (11.9)
  Day 7 | 1550 (11.4) | 1740 (19.7)

58. Primary Outcome: Cmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: Maximum observed plasma drug concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
nmol/L
  Day 1 | 738 (31.7)
  Day 7 | 1180 (33.2)

59. Primary Outcome: Tmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: Time to maximum plasma concentration was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 3.01 (32.7) [2.00 to 6.00] | 3.50 (27.9) [2.00 to 4.05] | 2.53 (62.7) [2.00 to 6.05] | 3.50 (37.7) [3.00 to 4.00] | 4.00 (63.2) [2.00 to 6.00]

60. Primary Outcome: Tmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
hours | 6.00 (48.5) [6.00 to 8.00]

61. Primary Outcome: Tmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
hours
  Day 1 | 3.00 (3.77) [2.00 to 3.05]
  Day 7 | 2.50 (21.7) [1.00 to 4.00]

62. Primary Outcome: Tmax of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
hours | 4.00 (39.8) [4.00 to 6.00] | 4.00 (49.1) [3.03 to 4.00] | 2.05 (20.4) [2.00 to 4.00] | 3.52 (NA) [3.03 to 4.00] | 4.00 (35.4) [1.00 to 6.00]

63. Primary Outcome: Tmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
hours
  Day 1 | 4.00 (51.4) [1.00 to 8.00] | 3.00 (52.9) [0.98 to 4.00] | 3.00 (45.4) [2.00 to 6.00] | 4.00 (40.1) [3.00 to 6.00]
  Day 7 | 2.00 (36.2) [1.92 to 6.00] | 2.00 (36.7) [1.00 to 3.00] | 3.00 (46.8) [1.00 to 4.00] | 4.00 (22.1) [2.00 to 4.00]

64. Primary Outcome: Tmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
hours
  Day 1 | 4.00 (51.7) [2.00 to 6.00] | 4.00 (45.0) [3.00 to 6.03]
  Day 7 | 4.00 (43.9) [2.00 to 4.00] | 4.00 (30.4) [3.00 to 6.00]

65. Primary Outcome: Tmax of M6 After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
hours | 4.00 (NA) [4.00 to 4.00]

66. Primary Outcome: Tmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1,HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
hours
  Day 1 | 3.00 (32.8) [2.00 to 4.00] | 4.00 (35.2) [3.00 to 4.00]
  Day 7 | 2.00 (31.8) [2.00 to 4.00] | 4.00 (23.2) [2.00 to 4.00]

67. Primary Outcome: Tmax of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: Time to maximum plasma concentration was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
hours
  Day 1 | 10.00 (44.0) [6.00 to 23.5]
  Day 7 | 4.00 (46.1) [3.00 to 8.00]

68. Primary Outcome: t1/2 of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Healthy Participants (Group A)
Description: as for outcome 33
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 22.5 (6.2) | 24.6 (12.8) | 29.1 (15.5) | 28.8 (14.2) | 22.9 (14.0)

69. Primary Outcome: t1/2 of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Fed State in Healthy Participants (Group A - Cohort 4a)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Uprifosbuvir 150 mg (Cohort 4a Fed)
Number analyzed (Participants) | 6
hours | 27.1 (9.1)

70. Primary Outcome: t1/2 of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Healthy Participants (Group A - Cohort 6a)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Uprifosbuvir 300 mg (Cohort 6a)
Number analyzed (Participants) | 6
hours | 32.2 (10.3)

71. Primary Outcome: t1/2 of M6 After Single Dose of Uprifosbuvir as the Capsule Formulation in Genotype 1, HCV-Infected Participants (Group B)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3
hours | 20.1 (3.4) | 21.2 (4.8) | 21.7 (19.8) | 26.9 (NA) — Not calculated | 28.0 (12.1)

72. Primary Outcome: t1/2 of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Capsule Formulation in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule)
Number analyzed (Participants) | 10 | 9 | 17 | 7
hours | 25.5 (16.8) | 28.9 (15.2) | 32.6 (12.7) | 35.8 (17.8)

73. Primary Outcome: t1/2 of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants (Group C)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group C: Uprifosbuvir 300 mg (Tablet) | Group C: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 7 | 7
hours | 32.4 (7.7) | 30.8 (26.8)

74. Primary Outcome: t1/2 of M6 After Single Dose of Uprifosbuvir as Capsule Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 1e)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group E: Uprifosbuvir 150 mg (Cohort 1e)
Number analyzed (Participants) | 2
hours | 24.0 (NA) — Not calculated

75. Primary Outcome: t1/2 of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as Capsule or Tablet Formulation in Genotype 1, HCV-Infected Participants With Mildly Impaired Hepatic Function (Child Pugh Class A) (Group E - Cohort 2e and Cohort 3e)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e)
Number analyzed (Participants) | 3 | 7
hours | 27.5 (9.3) | 26.2 (24.8)

76. Primary Outcome: t1/2 of M6 After Multiple Doses of Uprifosbuvir Once-Daily x 7 Days as the Tablet Formulation in Genotype 1, HCV-Infected Participants, With Itraconazole (Group F)
Description: The time measured for the plasma concentration to decrease by one half (t1/2) was obtained.
Time Frame: Days 1 & 7: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group F: Uprifosbuvir 300 mg (Tablet)
Number analyzed (Participants) | 8
hours | 38.9 (17.7)

77. Primary Outcome: Cumulative Urine Excretion of Unchanged Uprifosbuvir in Healthy Participants (Group A)
Description: Cumulative urine excretion of unchanged MK-3682 in healthy participants was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: umol
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
umol | 0.280 (0.0800) | 0.586 (0.164) | 7.73 (4.67) | 13.1 (4.16) | 1.56 (0.397)

78. Primary Outcome: Cumulative Urine Excretion of Unchanged M6 in Healthy Participants (Group A)
Description: Cumulative urine excretion of unchanged M6 in healthy participants was obtained. All participants were fasted.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: umol
Arm/Group | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 150 mg (Cohort 4a Fasted) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Uprifosbuvir 50 mg (Cohort 3a)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
umol | 5.93 (1.42) | 15.2 (2.50) | 101 (6.86) | 200 (37.9) | 31.8 (5.69)

79. Primary Outcome: Reduction in HCV RNA From Baseline on Day 8 Following Uprifosbuvir 50-450 mg for 7 Days in Genotype 1, 2 and 3, HCV-Infected Participants (Groups C and D)
Description: Reduction in HCV RNA from baseline on Day 8 following uprifosbuvir 50-450 mg for 7 Days in Genotype 1, 2 and 3, HCV-infected participants was obtained.
Time Frame: Baseline and Day 8
Population: Per-Protocol Population: participants who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Placebo (Pooled) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet)
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 8 | 7 | 7
log10 IU/mL
  Baseline | 5.82 (0.879) [1.00 to 8.00] | 6.00 (0.630) [0.98 to 4.00] | 6.16 (0.633) [2.00 to 6.00] | 6.11 (0.540) [3.00 to 6.00] | 6.27 (0.485) | 5.92 (0.838) | 5.97 (0.739)
  Day 8 | 0.78 (0.440) | 2.49 (0.733) | 4.22 (0.614) | 4.39 (0.433) | 0.42 (0.229) | 3.34 (0.643) | 4.50 (0.644)

80. Primary Outcome: Maximum Reduction in log10 HCV RNA From Baseline - Normal Participants (From Groups B and C) vs. Mild Hepatic Impairment Participants (Group E)
Description: Reduction in HCV RNA from baseline on Day 8 following uprifosbuvir 50-450 mg for 7 Days in Genotype (Gt) 1, HCV-infected participants was obtained.
Time Frame: Baseline and 28 days after last dose of study drug (Up to 42 days)
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Group C: Uprifosbuvir 300 mg (Capsule): Participants were administered single doses of uprifosbuvir 300 mg as oral capsules once daily for 7 days under fasted conditions.
- Group E: Uprifosbuvir 450 mg: Participants were administered single doses of uprifosbuvir 450 mg as oral tablets once daily for 7 days under fasted conditions.
Arm/Group | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group C: Uprifosbuvir 300 mg (Capsule) | Group E: Uprifosbuvir 450 mg
Number analyzed (Participants) | 2 | 8 | 7
log10 IU/mL
  Baseline | 5.91 (0.347) | 6.16 (0.633) | 6.14 (0.356)
  Normal hepatic fcn: Gt1a: number analyzed (Participants) | 1 | 3 | 2
  Normal hepatic fcn: Gt1a | 0.96 (NA) | 4.82 (0.504) | 5.06 (0.489)
  Mild hepatic impairment: Gt1a: number analyzed (Participants) | 0 | 2 | 1
  Mild hepatic impairment: Gt1a |  | 2.92 (0.239) | 3.60 (NA)
  Normal hepatic fcn: Gt1b: number analyzed (Participants) | 1 | 5 | 5
  Normal hepatic fcn: Gt1b | 1.35 (NA) | 3.82 (0.636) | 4.28 (0.584)
  Mild hepatic impairment: Gt1b: number analyzed (Participants) | 2 | 1 | 6
  Mild hepatic impairment: Gt1b | 1.36 (0.774) | 3.59 (NA) | 3.08 (1.06)
  Normal hepatic fcn: Gt1 (pooled 1a+1b) | 1.15 (0.274) | 4.19 (0.754) | 4.50 (0.644)
  Mild hepatic impairment;Gt1 (pooled 1a+1b): number analyzed (Participants) | 2 | 3 | 7
  Mild hepatic impairment;Gt1 (pooled 1a+1b) | 1.36 (0.774) | 3.15 (0.420) | 3.16 (0.989)

ADVERSE EVENTS:
Time Frame: Up to 42 days (28 days after last study drug administration)
Description: Safety Population: participants who received at least one dose of the study drug. For Cohort 4a, serious AEs and nonserious AEs are presented for participants on the fasted regimen.
Groups:
- Group A: Placebo (Cohort 1a - Cohort 5a - Pooled): Participants were administered a single dose of uprifosbuvir-matching placebo as oral capsules under fasted conditions (Cohorts 1a, 2a, 3a, 5a); Participants were administered single doses of uprifosbuvir-matching placebo as oral capsules on Days 1 and 7 in a 2-period crossover design (fasted/fed) with a 6 day washout between dosing periods (Cohort 4a).
Arm/Group | Group A: Placebo (Cohort 1a - Cohort 5a - Pooled) | Group A: Uprifosbuvir 10 mg (Cohort 1a) | Group A: Uprifosbuvir 25 mg (Cohort 2a) | Group A: Uprifosbuvir 50 mg (Cohort 3a) | Group A: Uprifosbuvir 150 mg (Cohort 4a) | Group A: Uprifosbuvir 300 mg (Cohort 5a) | Group A: Placebo (Cohort 6a) | Group A: Uprifosbuvir 300 mg (Cohort 6a) | Group B: Uprifosbuvir 10 mg (Cohort 1b) | Group B: Uprifosbuvir 25 mg (Cohort 2b) | Group B: Uprifosbuvir 50 mg (Cohort 3b) | Group B: Uprifosbuvir 150 mg (Cohort 4b) | Group B: Uprifosbuvir 300 mg (Cohort 5b) | Groups C & D: Uprifosbuvir 50 mg (Capsule) | Groups C & D: Uprifosbuvir 150 mg (Capsule) | Groups C & D: Uprifosbuvir 250 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Capsule) | Groups C & D: Uprifosbuvir 400 mg (Capsule) | Groups C & D: Uprifosbuvir 300 mg (Tablet) | Groups C & D: Uprifosbuvir 450 mg (Tablet) | Groups C & D: Placebo (Pooled) | Group E: Uprifosbuvir 150 mg (Cohort 1e) | Group E: Uprifosbuvir 300 mg (Cohort 2e) | Group E: Uprifosbuvir 450 mg (Cohort 3e) | Group F: Uprifosbuvir 300 mg (Tablet)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/11 | 0/10 | 0/8 | 0/18 | 0/8 | 0/8 | 0/8 | 0/9 | 0/3 | 0/3 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/10 | 0/6 | 2/6 | 2/6 | 4/6 | 3/6 | 1/2 | 2/6 | 1/3 | 2/3 | 1/3 | 2/3 | 2/3 | 8/11 | 7/10 | 7/8 | 8/18 | 5/8 | 6/8 | 5/8 | 6/9 | 0/3 | 3/3 | 5/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Placebo (Cohort 1a - Cohort 5a - Pooled) (N=10) | Group A: Uprifosbuvir 10 mg (Cohort 1a) (N=6) | Group A: Uprifosbuvir 25 mg (Cohort 2a) (N=6) | Group A: Uprifosbuvir 50 mg (Cohort 3a) (N=6) | Group A: Uprifosbuvir 150 mg (Cohort 4a) (N=6) | Group A: Uprifosbuvir 300 mg (Cohort 5a) (N=6) | Group A: Placebo (Cohort 6a) (N=2) | Group A: Uprifosbuvir 300 mg (Cohort 6a) (N=6) | Group B: Uprifosbuvir 10 mg (Cohort 1b) (N=3) | Group B: Uprifosbuvir 25 mg (Cohort 2b) (N=3) | Group B: Uprifosbuvir 50 mg (Cohort 3b) (N=3) | Group B: Uprifosbuvir 150 mg (Cohort 4b) (N=3) | Group B: Uprifosbuvir 300 mg (Cohort 5b) (N=3) | Groups C & D: Uprifosbuvir 50 mg (Capsule) (N=11) | Groups C & D: Uprifosbuvir 150 mg (Capsule) (N=10) | Groups C & D: Uprifosbuvir 250 mg (Capsule) (N=8) | Groups C & D: Uprifosbuvir 300 mg (Capsule) (N=18) | Groups C & D: Uprifosbuvir 400 mg (Capsule) (N=8) | Groups C & D: Uprifosbuvir 300 mg (Tablet) (N=8) | Groups C & D: Uprifosbuvir 450 mg (Tablet) (N=8) | Groups C & D: Placebo (Pooled) (N=9) | Group E: Uprifosbuvir 150 mg (Cohort 1e) (N=3) | Group E: Uprifosbuvir 300 mg (Cohort 2e) (N=3) | Group E: Uprifosbuvir 450 mg (Cohort 3e) (N=8) | Group F: Uprifosbuvir 300 mg (Tablet) (N=8)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site anaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 2 (4) | 4 (5) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator will submit any proposed publication to Sponsor for review and comment at least sixty (60) days prior to submission to a third party. If Sponsor believes in good faith that any proposed publication contains any proprietary or confidential information, Sponsor shall have the right to remove such references to such confidential information.